CLINICAL TRIAL: NCT03684889
Title: Pediatric and Young Adult Leukemia Adoptive Therapy (PLAT)-06: A Phase 1/2 Study of CD19-specific CAR T Cells With a Fully Human Binding Domain for CD19+ Leukemia or Lymphoma
Brief Title: CD19-specific CAR T Cells With a Fully Human Binding Domain for CD19+ Leukemia or Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-06
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Leukemia; Lymphoma
Keywords: CAR T cell, CD19, pediatric, young adults
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCRI-huCAR19v2 (Experimental): Patients will receive SCRI-huCAR19v2 in either Phase 1 or Phase II
  Interventions: Biological: SCRI-huCAR19v2
- SCRI-huCAR19v1 - [CLOSED] (Experimental): Patients will receive SCRI-huCAR19v1 in either Phase 1 or Phase II. As of 02/13/2020 this study cohort is permanently closed.
  Interventions: Biological: SCRI-huCAR19v1

INTERVENTIONS:
Biological: SCRI-huCAR19v1 — 1:1 mixture of CD4:CD8 autologous T cells lentivirally transduced to express a second generation 4-1BB-ζ human CD19-specific CAR and Her2tG
  Arms: SCRI-huCAR19v1 - [CLOSED]
Biological: SCRI-huCAR19v2 — Mixture of CD4:CD8 autologous T cells lentivirally transduced to express a second generation 4-1BB-ζ human CD19-specific CAR and Her2tG
  Arms: SCRI-huCAR19v2

SUMMARY:
Patients with relapsed or refractory leukemia or lymphoma are often refractory to further chemotherapy. In this study, the investigators will attempt to use T cells obtained directly from the patient, which can be genetically engineered to express a fully human chimeric antigen receptor (CAR). The CAR used in this study can recognize CD19, a protein expressed on the surface of leukemia and lymphoma cells. The fully human CAR used in this study may help protect against rejection of the CAR T cells, which in turn could lead to lasting protection against return of the leukemia or lymphoma. The phase 1 part of this study will determine the safety of these CAR T cells, and the phase 2 part of the study will determine how effective this CAR T cell therapy is. Both patients who have never had prior CAR T cell therapy and those who have had prior CAR T cell therapy may be eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age ≥ 1 and ≤ 30 years
* First 2 enrolled subjects: age ≥ 18 and ≤ 30 years
* Disease requirements:

  * Phase 1: Evidence of refractory or recurrent CD19+ leukemia or lymphoma following previous CAR T cell immunotherapy
  * Phase 2: Evidence of refractory or recurrent CD19+ leukemia or lymphoma
* Able to tolerate apheresis, or has sufficient existing apheresis product or T cells for manufacturing investigational product
* Life expectancy ≥ 8 weeks
* Lansky or Karnofsky, as applicable, score ≥ 50
* Recovered from acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy, if the subject does not have a previously obtained apheresis product that is acceptable and available for manufacturing of CAR T cells
* ≥ 7 days post last chemotherapy and biologic therapy, with the exception of intrathecal chemotherapy and maintenance chemotherapy
* No prior virotherapy
* ≥ 7 days post last corticosteroid therapy
* ≥ 3 days post Tyrosine Kinase Inhibitor (TKI) use
* ≥ 1 day post hydroxyurea
* 30 days post most recent CAR T cell infusion
* Adequate organ function
* Adequate laboratory values, including absolute lymphocyte count ≥ 100 cells/uL
* Subjects of childbearing or child-fathering potential must agree to use highly effective contraception from consent through 12 months following infusion of investigational product on trial
* Subject and/or legally authorized representative has signed the informed consent form for this study

Exclusion Criteria:

* Presence of active malignancy other than disease under study
* History of symptomatic CNS pathology or ongoing symptomatic CNS pathology
* CNS involvement of leukemia or lymphoma that is symptomatic and in the opinion of the investigator, cannot be controlled during the interval between enrollment and CAR T cell infusion
* Presence of active GVHD, or receiving immunosuppressive therapy for treatment or prevention of GVHD within 4 weeks prior to enrollment
* Presence of active severe infection
* Presence of primary immunodeficiency syndrome
* Subject has received prior virotherapy
* Pregnant or breastfeeding
* Subject and/or legally authorized representative unwilling to provide consent/assent for participation in the 15-year follow up period, required if CAR T cell therapy is administered
* Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with CAR T cell product infusions will be assessed | 30 days
  The type, frequency, severity, and duration of adverse events will be summarized
The leukemia response to SCRI-huCAR19 in subjects with relapsed or refractory CD19+ leukemia will be assessed | 63 days
  Response will be defined by standard bone marrow assessment and standard response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, MD, Study Chair — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No